CLINICAL TRIAL: NCT01964547
Title: A Multicentre, Double-blind, Randomised, Parallel Group, Placebo-controlled Study of the Effect of Long-term Treatment With Sativex on Cognitive Function and Mood of Patients With Spasticity Due to Multiple Sclerosis
Brief Title: A Randomized Study of Sativex on Cognitive Function and Mood: Multiple Sclerosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWMS1137
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis; Spasticity
Keywords: Cognition; Mood
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Active Comparator): Contains delta-9-tetrahydrocannabinol (THC), 27 mg/mL:cannabidiol (CBD), 25 mg/mL, in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Each actuation delivers THC 2.7 mg and CBD 2.5 mg.
  Dose: 100 µL oromucosal spray to be administered up to a maximum of 12 sprays per day. There was an initial dose-titration period during which patients gradually increased their dose of study drug according to individual response and tolerability.
  Interventions: Drug: Sativex
- Placebo (Placebo Comparator): Oromucosal spray, containing ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring and colourings FD&C Yellow No.5 (E102 tartrazine) (0.0260%), FD&C Yellow No.6 (E110 sunset yellow) (0.0038%), FD&C Red No. 40 (E129 Allura red AC) (0.00330%) and FD&C Blue No.1 (E133 Brilliant blue FCF) (0.00058%). Dose: 100 µL oromucosal spray to be administered up to a maximum of 12 sprays per day. There was an initial dose-titration period during which patients gradually increased their dose of study drug according to individual response and tolerability.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — Patients self-administered their allocated randomized treatment on an outpatient basis, up to a maximum of 12 sprays to the oral mucosa per day (following an initial titration period).
  Other Names: Nabiximols; GWP42001; THC/CBD spray
  Arms: Sativex
Drug: Placebo — Patients self-administered their allocated randomized treatment on an outpatient basis, up to a maximum of 12 sprays to the oral mucosa per day (following an initial titration period).
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
A study to compare the change in cognitive performance and psychological status of patients with spasticity due to Multiple Sclerosis when treated with Sativex or placebo, added to existing anti-spasticity therapy over a period of 48 weeks. Secondary objectives were to evaluate the effect of Sativex on mood and spasticity and to assess the safety and tolerability of Sativex.

DETAILED DESCRIPTION:
Eligible patients entered this 50 week multicenter, double-blind, randomised, placebo-controlled, parallel group study which evaluated the effect of Sativex on cognitive performance. At each scheduled clinic visit, patients were assessed for cognitive performance, mood, severity of spasticity, use of investigational medicinal products and number of visits to a healthcare professional. Primary efficacy comparisons were made between scores recorded during baseline and scores recorded at the end of treatment.

ELIGIBILITY:
Inclusion Criteria (ALL to be fulfilled):

* Patient is willing and able to give informed consent for participation in the study.
* Patient is aged 18 years or above.
* Diagnosed with any disease sub-type of multiple sclerosis.
* Diagnosed with symptomatic spasticity due to multiple sclerosis.
* Patient has at least moderate spasticity in the opinion of the investigator.
* Patient fulfils at least one of the two criteria below. Subject must be either:

  * Currently established on a regular dose of anti-spasticity therapy, or
  * Previously tried and failed anti-spasticity therapy.
* Stable medication regimen for at least four weeks prior to study entry, for all medications which may have an effect on spasticity and/or cognition.
* If the patient is taking disease modifying medication this must be at a stable dose for three months prior to the initial visit.
* Willing and able to comply with all study requirements.
* Willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable.
* Willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria (if ANY apply):

* Any history or immediate family of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Any concomitant disease or disorder (such as poorly controlled epilepsy or seizures) that may influence the patient's level of cognition or mood.
* Currently using or has used cannabis or cannabinoid-based medications within 30 days of study entry and unwilling to abstain for the duration of the study.
* Any known or suspected history of a diagnosed dependence disorder, current heavy alcohol consumption (more than 60g of pure alcohol per day for men, and more than 40g of pure alcohol per day for women), current use of an illicit drug or current non-prescribed use of any prescription drug.
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal products.
* Female patients of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
* Female patient who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Patients who have received an investigational medicinal product within the 12 weeks prior to the initial visit.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study may influence the result of the study, or the patient's ability to participate in the study.
* Following a physical examination, the patient has any abnormalities that, in the opinion of the investigator would prevent the patient from safe participation in the study.
* Previously randomised to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MS Centre, Charles University, Prague, Czechia

REFERENCES:
- [Result] Abstracts of ECTRIMS (Congress of the European Committee for Treatment and Research in Multiple Sclerosis) 2013. October 2-5, 2013. Copenhagen, Denmark. Mult Scler. 2013 Oct;19(11 Suppl):8-597. No abstract available. PMID 24151639
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Each 100 μl actuation contains delta-9-tetrahydrocannabinol (THC) (27 mg/mL) and CBD (25 mg/mL). The maximum permitted dose was 12 actuations (32.4 mg THC + 30 mg CBD) in any 24 hour period.
- Placebo: Each 100 μl actuation contains no active drug but colorants and excipients. The maximum permitted dose was 12 actuations in any 24 hour period.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 62 | 59
Completed | 50 | 48
Not Completed | 12 | 11
Not completed — Adverse Event | 8 | 2
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Investigator | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sativex: Each 100 μl actuation contains THC (27 mg/mL) and CBD (25 mg/mL). The maximum permitted dose was 12 actuations (32.4 mg THC + 30 mg CBD) in any 24 hour period.
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 58 | 119
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.95 (8.954) | 48.21 (10.381) | 48.59 (9.642)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 23 | 22 | 45
Region of Enrollment [Number; unit: participants]
  Czech Republic | 62 | 59 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of Treatment in Paced Auditory Serial Addition Test (PASAT) Total Score.
Description: The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. Stimulus presentation rates were adapted for use with multiple sclerosis patients. The PASAT is presented on audio compact disk to control the rate of stimulus presentation. Single digits are presented either every 3 seconds (PASAT 1) or every 2 seconds (PASAT 2), and the patient must add each new digit to the one immediately prior to it. The test score is the sum of the total number of correct sums given (out of 60 possible) in each trial. An increase in score indicates an improvement in condition.
Time Frame: 0-48 weeks
Population: All randomized patients who received at least one dose of study medication and yielded on-treatment efficacy data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 55 | 52
units on a scale | 6.8 (16.16) | 6.8 (13.49)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change at end of treatment was compared between treatment groups using ANCOVA. The model included treatment group and center grouping as factors and the baseline score as covariate. The planned sample size was 120 participants(60 patients in the Sativex arm and 60 in the placebo arm); Test type: Non-Inferiority or Equivalence — The sample size is adequate to confirm the non-inferiority of Sativex with a clinical relevant reduction delta of 10%, assuming there is no difference between treatments in the actual change in cognition and also assuming a standard deviation for treatment difference of 10, using a one-tailed 2.5% significance level and power of 90%. Sativex is deemed to be non-inferior to placebo if the lower 1-sided 97.5% CI of the estimated mean treatment difference (Sativex-Placebo) is greater than -10%; ANCOVA; Estimated mean treatment difference = -1.47, 97.5% CI 1-sided [lower limit -6.41], Standard Error of Mean 2.492

2. Secondary Outcome: Change From Baseline to the End of Treatment in Beck Depression Inventory-II (BDI-II) Total Score.
Description: The BDI-II is a multiple choice self-reported inventory that is one of the most widely used instruments for measuring the severity of depression. There are 21 questions or items, each having four possible responses. Each response is assigned a score ranging from zero to three, indicating the severity of the symptom. Items 1 to 13 assess symptoms that are psychological in nature, while items 14 to 21 assess symptoms that are more physical. The sum of all BDI-II item scores indicates the severity of depression. For patients eligible for this study, a score of 21 or over represents depression. The BDI-II can distinguish between different subtypes of depressive disorders, such as major depression and dysthymia. A reduction in score indicates an improvement in condition.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 57 | 56
units on a scale | -3.1 (7.76) | -2.4 (6.38)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change at end of treatment was compared between treatment groups using ANCOVA. The model included treatment group and center grouping as factors and the baseline score as covariate; Test type: Non-Inferiority or Equivalence — Sativex is deemed to be non-inferior to placebo if the upper 1-sided 97.5% CI of the estimated mean treatment difference (Sativex-Placebo) is less than +5%; ANCOVA; Estimated mean treatment difference = -0.29, 97.5% CI 1-sided [upper limit 2.33], Standard Error of Mean 1.323

3. Secondary Outcome: Subject Global Impression of Change (SGIC) in the Severity of Their Spasticity at the End of Treatment.
Description: Patients were asked the following question, to be rated on a seven-point scale:
  "Please assess the change in your spasticity since immediately before receiving the first dose of study treatment (Visit 1) using the scale below".
  The markers were: 'Very much worse', 'Much worse', 'Minimally worse', 'No change', 'Minimally better', 'Much better' or 'Very much better'.
  The number of patients for each of the markers is presented at the final study visit.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 58 | 56
participants
  Very Much Better | 2 | 0
  Much Better | 16 | 6
  Minimally Better | 24 | 15
  No Change | 13 | 27
  Minimally Worse | 1 | 7
  Much Worse | 2 | 1
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Sativex vs Placebo; Data were analysed using ordinal logistic regression using the cumulative proportional odds model, with global impression of change as the dependent variable and treatment group as factor; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.02, 95% CI 2-sided [1.96 to 8.22]

4. Secondary Outcome: Caregiver's Global Impression of Change (CGIC) in the Severity of the Patient's Spasticity at the End of Treatment.
Description: Caregivers were asked the following question to be rated on a seven-point scale:
  "How has the subject's spasticity changed since Visit 1?" The markers were: Very much worse, Much worse, Minimally worse, No change, Minimally better, Much better, Very much better.
  The number of patients for each of the markers is presented at the final study visit.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 41 | 40
participants
  Very Much Better | 1 | 0
  Much Better | 12 | 6
  Minimally Better | 14 | 10
  No Change | 11 | 18
  Minimally Worse | 3 | 3
  Much Worse | 0 | 3
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0142, Regression, Logistic; Odds Ratio (OR) = 2.79, 95% CI 2-sided [1.23 to 6.31]

5. Secondary Outcome: Physician's Global Impression of Change (PGIC) in the Severity of the Patient's Spasticity at the End of Treatment.
Description: Physicians were asked the following question to be rated on a seven-point scale:
  "How has the subject's spasticity changed since Visit 1?" The markers were: Very much worse, Much worse, Minimally worse, No change, Minimally better, Much better, Very much better.
  The number of patients for each of the markers is presented at the final study visit.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 58 | 56
participants
  Very Much Better | 0 | 1
  Much Better | 15 | 6
  Minimally Better | 26 | 15
  No Change | 14 | 29
  Minimally Worse | 3 | 4
  Much Worse | 0 | 1
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 3.07, 95% CI 2-sided [1.51 to 6.21]

6. Secondary Outcome: Change From Baseline to End of Treatment in Modified Ashworth Scale Total Score.
Description: All 20 muscle groups were assessed for spasticity (using a 0-5 scale): 0= 'no increase in muscle tone' to 5= 'affected part(s) rigid in flexion or extension'. The score for all 20 muscle groups were added to give a total score out of 100. A decrease in score indicates an improvement in condition.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 58 | 56
units on a scale | -10.6 (11.26) | -7.7 (10.70)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.212, ANCOVA; Estimated mean treatment difference = -2.36, 95% CI 2-sided [-6.09 to 1.37], Standard Error of Mean 1.880

7. Secondary Outcome: Change From Baseline to End of Treatment in Number of Visits to a Healthcare Professional.
Description: At baseline, patients were asked how many times they had visited a healthcare professional in the previous 12 weeks. At subsequent visits, patients were asked how many times they had visited a healthcare professional since their last study visit. The change from baseline to the end of treatment is presented. A decrease in number indicates an improvement in condition.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 58 | 56
visits | -0.6 (0.99) | -0.4 (1.30)

8. Secondary Outcome: The Number of Patients With a Treatment-emergent Flag Using the Columbia-Suicide Severity Rating Scale (C-SSRS) During the Course of the Study.
Description: Patients were scored at each clinic visit for the following outcomes using the C-SSRS: suicidal ideation, suicidal behaviour, suicidality (including complete suicidality). Possible flags were as follows: "Wish to be Dead", "Non-specific Active Suicidal Thoughts", "Active Suicidal Ideation Without Intent", "Active Suicidal Ideation With Intent, No Plan", "Active Suicidal Ideation With Intent and Plan". The number of patients with a treatment-emergent flag is presented.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 62 | 59
participants
  Wish to be Dead | 0 | 2
  Non-specific Active Suicidal Thoughts | 0 | 1
  Active Suicidal Ideation Without Intent | 0 | 1
  Active Suicidal Ideation With Intent, No Plan | 0 | 0
  Active Suicidal Ideation With Intent and Plan | 0 | 0

9. Secondary Outcome: Change From Baseline to End of Treatment in Timed 10-meter Walk Times.
Description: Only those patients for whom it was appropriate (i.e. ambulatory patients) were timed for how long it took to walk 10 metres. If a patient started the 10-meter walk but was unable to complete it, an estimated time for completion was calculated based on the available data. A negative difference from baseline indicates an improvement in condition.
Time Frame: 0-48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 47 | 50
seconds | 6.2 (55.34) | 3.0 (24.68)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change at end of treatment was compared between treatment groups using ANCOVA. The model included treatment group and centre grouping as factors and baseline score as covariate; Test type: Superiority or Other; p = 0.556, ANCOVA; Estimated mean treatment difference = 4.88, 95% CI 2-sided [-11.51 to 21.27], Standard Error of Mean 8.250
Statistical Analysis 2: Comparison: Sativex vs Placebo; The change at end of treatment was compared between treatment groups using non-parametric methods as the distribution of data was non-normal; Test type: Superiority or Other; p = 0.088, Wilcoxon (Mann-Whitney); Hodges-Lehmann median difference = -1, 95% CI 2-sided [-3 to 0]

10. Secondary Outcome: Incidence of Adverse Events as a Measure of Patient Safety.
Description: The number of subjects who experienced an adverse event during the course of the study is presented.
Time Frame: 0-50 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 62 | 59
participants | 39 | 19

ADVERSE EVENTS:
Time Frame: All adverse events occurring during the study (0-50 weeks) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 5/62 | 0/59
Other Adverse Events (participants affected / at risk) | 34/62 | 19/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=62) | Placebo (N=59)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 — The acute myocardial infarction resulted in the affected participant's death; this was not considered to be treatment-related.
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Drug Withdrawal Syndrome (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=62) | Placebo (N=59)
Vertigo (Ear and labyrinth disorders) | 6 | 0
Visual Impairment (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Oral Mucosal Erythema (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 5 | 1
Pyrexia (General disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Bacterial Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 5 | 1
Viral Infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Face Injury (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1
Vitamin D Decreased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebellar Ataxia (Nervous system disorders) | 2 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 1 | 2
Memory Impairment (Nervous system disorders) | 1 | 0
Multiple Sclerosis (Nervous system disorders) | 1 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 3 | 4
Muscle Spasticity (Nervous system disorders) | 5 | 2
Neuralgia (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Stupor (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Trigeminal Neuralgia (Nervous system disorders) | 1 | 0
Anxiety Disorder Due To A General Medical Condition (Psychiatric disorders) | 2 | 0
Euphoric Mood (Psychiatric disorders) | 2 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal Blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Lipoma Excision (Surgical and medical procedures) | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 1 | 0
Application Site Discomfort (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW Pharma Ltd (GW) will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.